CLINICAL TRIAL: NCT00003023
Title: Phase I Trial of A1G4 Anti-Idiotypic Monoclonal Antibody With Bacille-Calmette-Guerin (BCG) Adjuvant in High Risk Patients With GD2 Positive Tumors
Brief Title: Monoclonal Antibody A1G4 Plus BCG in Treating Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-024; P30CA008748 (NIH); MSKCC-97024; NCI-G97-1268
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Neuroblastoma; Sarcoma
Keywords: metastatic osteosarcoma; recurrent adult soft tissue sarcoma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; recurrent osteosarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Osteosarcoma | interventions — BCG Vaccine

INTERVENTIONS:
Biological: BCG vaccine
Biological: monoclonal antibody A1G4 anti-idiotype vaccine

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody A1G4 with BCG may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody A1G4 plus BCG in treating patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the toxicity and feasibility of immunizing patients with anti-idiotypic rat monoclonal antibody A1G4 combined with Bacillus Calmette Guerin (BCG) adjuvant.
* Determine whether immunization with A1G4 combined with BCG results in an immune response directed against GD2 ganglioside in patients.

OUTLINE: All patients are treated with A1G4 diluted in sterile physiologic saline mixed with Bacillus Calmette Guerin (BCG) organisms. The vaccine is injected intradermally in multiple sites. Booster immunizations are administered during weeks 2, 4, 8, 12, 20, 28, 36, 44, 52. Immunizations are not administered in limbs where draining lymph nodes have been surgically removed or previously irradiated. Isoniazid is administered for 5 days after each BCG injection. If severe skin reactions are present at the injection site, the BCG dose is decreased. If skin reactions persist, the BCG dose is stopped but A1G4 injections continue.

At least 6 patients are accrued at each dose level of A1G4. Dose escalation is not carried out until patients have been followed for at least 8 weeks after the first immunization without encountering grade 3 or worse non-skin toxicity.

If 0-1 patient experiences dose limiting toxicity (DLT) at a given dose level, then patients are accrued to the next higher dose level. If 2 or more patients experience DLT, the MTD is defined as the previous dose level.

Patients are followed for at least 1 year.

PROJECTED ACCRUAL: A total of 24 patients are expected to complete this study. If patients are removed early from the study prior to evaluation for serological response, additional patients will be accrued until 6 patients are evaluable for serological response.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed GD2 positive tumors which include:

  * High risk neuroblastoma (stage IV, or N-myc amplified, or localized neuroblastoma multiply recurrent)
  * Recurrent or metastatic osteosarcoma
  * Recurrent or metastatic GD2 positive sarcomas
* If free of disease, patient must be fully recovered from toxic effects or complications of prior treatments (chemotherapy or surgery)

  * No greater than 6 months since last chemotherapy or surgery before first injection of A1G4

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* At least 6 months

Hematopoietic:

* Absolute neutrophil count greater than 500/mm^3
* Absolute leukocyte count greater than 500/mm^3
* Peripheral T-cell phytohemagglutinin activation (PHA) at least 50% of normal

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No significant heart disease (NYHA class III or IV)

Other:

* No other serious intercurrent illnesses
* No active infections requiring antibiotics
* No active bleeding
* No primary immunodeficiency
* Not pregnant or nursing
* Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent antibiotics
* No prior mouse antibodies and detectable human antimouse antibody (HAMA) titer

Chemotherapy:

* See Disease Characteristics
* At least 6 weeks since nitrosoureas
* At least 4 weeks since other systemic chemotherapy

Endocrine therapy:

* No concurrent nonsteroidal anti-inflammatory agents
* No concurrent corticosteroid

Radiotherapy:

* At least 4 weeks since radiotherapy
* No prior radiation therapy to the spleen

Surgery:

* See Disease Characteristics
* No splenectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1997-03; Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong V. Cheung, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States